CLINICAL TRIAL: NCT01738607
Title: The Impact of Fiber Fermentation on Fecal Incontinence
Brief Title: Dietary Fiber for Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 010M69241; R01NR007756-01A2 (NIH)
Record Dates: First submitted 2012-11-21; First posted 2012-11-30 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence, dietary fiber
MeSH Terms: conditions — Fecal Incontinence | interventions — Psyllium; Gum Arabic; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): basic recipe for juice and muffin recipe
  abbreviated PLB
  Interventions: Dietary Supplement: Placebo
- Carboxymethylcellulose (Experimental): The supplements were prepared as two fruit juice mixtures (each 270 ml) providing 7 g total fiber/d) and two small muffins providing 9 g total fiber/d for 16 g of toal fiber daily.
  abbreviated CMC
  Interventions: Dietary Supplement: carboxymethylcellulose
- Gum Arabic (Experimental): The supplements were prepared as two fruit juice mixtures (each 270 ml) providing 7 g total fiber/d) and two small muffins providing 9 g total fiber/d for 16 g of toal fiber daily.
  abbreviated GA
  Interventions: Dietary Supplement: Gum Arabic
- Psyllium (Experimental): The supplements were prepared as two fruit juice mixtures (each 270 ml) providing 7 g total fiber/d) and two small muffins providing 9 g total fiber/d for 16 g of toal fiber daily.
  abbreviated as PSY
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Dietary Supplement: Psyllium
  Arms: Psyllium
Dietary Supplement: Gum Arabic — Gum acacia dietary fiber
  Other Names: Gum acacia
  Arms: Gum Arabic
Dietary Supplement: carboxymethylcellulose — dietary fiber
  Arms: Carboxymethylcellulose
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The primary aim of this study was to compare the effects of supplementation with one of three dietary fibers (gum arabic, carboxy-methylcellulose, or psyllium) or a placebo on fecal incontinence (FI), symptom intolerance, and quality of life in community-living individuals who have incontinence of loose or liquid feces. A secondary aim was to explore the possible mechanism(s) underlying the supplements' efficacy (i.e., improvements in stool consistency, water-holding capacity or gel formation).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* living in the community (not a nursing home or assisted living facility)
* self-report of usually having FI of loose or liquid consistency at least twice in a 2-wk period
* toilets independently
* ability to read and write in English.
* Persons that regularly performed pelvic floor muscle exercises and/or biofeedback on a maintenance regimen for at least 20 wks or who took a steady dose of anti-motility medications on a regular schedule that still met the FI criteria were also eligible.

Exclusion Criteria:

* difficulty swallowing,
* a gastrointestinal (GI) tract altered by surgery,
* a malabsorption disorder,
* inflammatory bowel disease,
* gastrointestinal cancer or active cancer treatment,
* allergy to the fibers,
* regularly used a laxative or enema, were tube-fed, or unwilling to discontinue taking periodic self-prescribed fiber supplements or anti-diarrheal medications.
* a score ≤24 on the Mini Mental State Examination
* having/reporting fewer than two episodes of FI or being incapable of performing study procedures during the run-in baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2004-04; Primary Completion 2007-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
self-report of an incontinent episode on a daily stool diary
  the date and time of an incontinence episode was reported and the ratio of the number of incontinence episodes to total stools daily was calculated

SECONDARY OUTCOMES:
self-report of gastro-intestinal symptoms on a daily symptom record
  The amount of GI symptoms reported were flatus, belching, bloating, abdominal cramping, nausea, a feeling of fullness, and stomach upset using a categorical scale. Number of times of flatus was also reported.
  The amount of two obfuscating symptoms were also reported. headache and sleepiness.
  How upsetting/bothersome the symptoms were were also reported.
self-report of quality of life
  The Fecal Incontinence Quality of Life tool (FIQL) was used; Rockwood, T.H. et al. Diseases of the Colon & Rectum. 2000;43(1):9-16.
Water-holding capacity of non-frozen of stools
  Measure was done on stools of 52 randomly selected subjects (13 from each group) Established method of Wenzl, H. et al. Gastroenterology. 1995;108(6):1729-38 used.
Gel formation of non-frozen stools
  Measure was done on stools of 52 randomly selected subjects (13 from each group); Established method of Fischer, M.H. et al.Carbohydrate Research 2004;339(11): 2009-2017.
Total dietary fiber content of feces
  Measured in composites of all stools from baseline and supplement periods and non-frozen stools
  Established method of Theander O, et al. J AOAC Int. 1995;78(4):1030-44 used.
Self-report of amount of supplement consumed
  reported by fractions on supplement intake form and return of unconsumed portion was assessed by study team
amount of fecal incontinence
  subjects self-reported greatest amount of soiling (from soling of tissue between buttocks to shoes or floor)
wet and dry weights of collected stools and percentage of water content
  collected stools were weighed and freeze-dried to constant weight; percentage of water content was calculated from these values

OTHER OUTCOMES:
self-reported rating of consistency of continent stools on a daily stool diary
  the Stool Consistency Classification System used was shown to be valid and reliable
usual diet intake
  written record of all food and drink consumed
report of additional fluid intake
  subjects checked whether the drank required amount of additional fluid and wrote the date and time of drinking
absorbent pad soiling
  subjects indicated number of absorbent products that were soiled on stool diary and and saved and returned them to be assessed by study team
self-report of any stools not collected
  reported on stool diary daily with reason for not collecting
Stool Color change
  date and time a stool color change was observed after swallowing a capsule with a decoy or marker dose of a food dye; date and time capsule was taken was also reported
in vitro fiber degradation
  nested experiment of in vitro degradation of each dietary fiber by stools of subjects using established procedure reported in Bliss, D.Z. et al. Nurs. Res. 2001, 50, 203-213.
total dietary fiber content of fiber sources used in Study
  established method of Theander O. et al. J AOAC Int. 1995;78(4):1030-44 used.
Personal Goals of Treatment for Fecal Incontinence and Satisfaction with Achievement of Goals
  data obtained by semi-structured interview
modifications of preparation of foods, diet intake, and eating pattern to manage fecal incontinence
  data obtained by semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Donna Z Bliss, phD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States